CLINICAL TRIAL: NCT06893835
Title: Comparative Study of Clinical Outcomes and Safety Between Colistin and Tigecycline for Multi-Drug Resistant Gram Negative Bacteria
Brief Title: Comparative Study of Clinical Outcomes and Safety Between Colistin and Tigecycline
Acronym: MDRS
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Nada Abd El-Hamed Saad Rezk, Pharmacist, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Multidrug resistance
Record Dates: First submitted 2025-03-06; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-02

CONDITIONS: Infection in ICU
Keywords: colistin; Tigecycline; renal impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — colistinmethanesulfonic acid; Colistin; Tigecycline

STUDY DESIGN:
Intervention Model Description: Group I: 66 patients received intravenous colistin 300 mg colistin base activity (CBA) as loading dose, followed by 2.5-5mg/kg/day of CBA in 2 divided doses as a maintenance dose in intensive care unit to treat their MDR infection.
  Group II: 66 patients received intravenous tigecycline100 mg single dose as loading dose, followed by 25-50 mg every 12 hours maintenance dose in intensive care unit to treat their MDR infection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Colistin (Active Comparator): Intravenous colistin 300 mg colistin base activity (CBA) as loading dose, followed by 2.5-5mg/kg/day of CBA in 2 divided doses as a maintenance dose.
  Reconstitute each vial of CBA with 2 ml of sterile water for injection, swirl gently. further dilute in normal saline.
  Interventions: Drug: Colistimethate Sodium
- Tigecycline (Active Comparator): intravenous tigecycline100 mg single dose as loading dose, followed by 25-50 mg every 12 hours maintenance dose.
  add 5.3 ml normal saline to each 50 ml vial. swirl gently. further dilution to final concentration does not exceed 1mg/ml.
  Interventions: Drug: Tigecycline

INTERVENTIONS:
Drug: Colistimethate Sodium — compare the clinical outcomes and safety between colistin and tigecycline for multi-drug-resistant gram-negative bacteria.
  Other Names: colistin
  Arms: Colistin
Drug: Tigecycline — compare the clinical outcomes and safety between colistin and tigecycline for multi-drug-resistant gram-negative bacteria.
  Other Names: tygcil
  Arms: Tigecycline

SUMMARY:
Objective from this study to compare the clinical outcomes and safety between colistin and tigecycline for multi-drug resistant gram negative bacteria.

DETAILED DESCRIPTION:
Study will be in Beni-Suef university hospital. Group I: 66 patients received intravenous colistin 300 mg colistin base activity (CBA) as loading dose, followed by 2.5-5mg/kg/day of CBA in 2 divided doses as a maintenance dose in intensive care unit to treat their MDR infection and group 2 contains 66 patients received intravenous tigecycline100 mg single dose as loading dose, followed by 25-50 mg every 12 hours maintenance dose in intensive care unit to treat their MDR infection

ELIGIBILITY:
Inclusion criteria:

Study will include

* adult patient (male, female)
* age from 18 to 70 years
* Patients admitted to intensive care unit in study period (six months) who received intravenous colistin or tigecycline as antimicrobial drug for treatment their MDR gram negative infection.

Exclusion criteria:

* Patient admitted to intensive care unit younger than 18 years or older than 70 years.
* Liver transplantation patients.
* Patients are chronic kidney disease (CKD on hemodialysis or baseline creatinine clearance (crcl) < 10 ml/min (estimated by Cockcroft Gault equation).
* Patients received renal replacement therapy before or during admission.
* Patient is on any other nephrotoxic drug (vancomycin, aminoglycosides, NSAIDs, cyclosporine, amphotericin B, etc.).
* Pregnant and lactating women.
* Patients refused the consent of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
comparison clinical success between colistin and tigecycline | 6 months
  the disappearance of clinical signs and symptoms as normalization of leukocyte counts and resolution of fever after receiving colistin and tigecycline

CONTACTS AND LOCATIONS:
Overall Officials: Shimaa N Abd elfatah, PhD, Study Chair — Beni-Suef University
Locations (1):
- Pharmacy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2024-11-01): https://cdn.clinicaltrials.gov/large-docs/35/NCT06893835/Prot_000.pdf